CLINICAL TRIAL: NCT06141954
Title: Therapeutic Ultrasound Versus Low Level Laser Therapy on Postpartum Sacroiliac Joint Pain
Brief Title: US vs Low Level Laser on Sacroiliac Postpartum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Ibrahim Seif Eldein, physiotherapy practitioner, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: US vs Low level laser
Record Dates: First submitted 2023-11-09; First posted 2023-11-21 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Sacroiliac Disorder
Keywords: Ultrasound therapy; Low level laser therapy
MeSH Terms: interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: Comparison between effect of ultrasound and low level laser on sacroiliac joint pain in woman postpartum
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound (Active Comparator): Effect of ultrasound therapy on sacroiliac joint pain in woman postpartum
  Interventions: Device: Ultrasound waves therapy
- Low level laser (Active Comparator): Effect of low level laser therapy on sacroiliac joint pain in woman postpartum
  Interventions: Device: Low level laser therapy

INTERVENTIONS:
Device: Ultrasound waves therapy — Therapeutic ultrasound is proposed to deliver energy to deep tissue sites through ultrasonic waves, to produce increases in tissue temperature or non- thermal physiologic changes. Low level laser therapy penetrates particularly light waves that increase cellular metabolism.
  Arms: Ultrasound
Device: Low level laser therapy — Low-level laser (light) therapy (LLLT) is a fast-growing technology used to treat a multitude of conditions that require stimulation of healing, relief of pain and inflammation, and restoration of function.
  Arms: Low level laser

SUMMARY:
This study will be conducted to compare between effect of therapeutic ultrasound and low-level laser therapy on sacroiliac joint pain after delivery.

DETAILED DESCRIPTION:
Women are more prone to sacroiliac joint (SIJ) pain during pregnancy and after childbirth. The hormonal changes during pregnancy and lactation make all the ligaments of the woman's body more lax and more flexible. Also, these hormones increase mobility of SIJs that are usually pretty stable, this in turn can leave the SIJs too mobile and can cause inflammation and pain in SIJ. In general, women are 8 to 10 times likely to experience SIJ pain and dysfunction than men due to the differences in their anatomy and body chemistry. Also, some studies have shown that, the younger woman has a greater risk of developing SIJ pain than the older one.On the other hand, the incidence of SIJ pain after delivery is very high and is more than we might think, since about 15-30% of postpartum women have SIJ pain. The pain starts when the mother's SIJs get inflamed. The SIJ pain can increase risk of low back pain after delivery.

The main cause of SIJ pain after delivery is the hypermobility and instability of SIJs. Hypermobility of SIJs caused by the pregnancy hormones causes an alteration in the normal joint motion (too much movement) which in turn causes instability in SIJs. About 30% of SIJ patients have postpartum instability in their SIJs so, they experience SIJ pain after delivery.Core weakness or muscle imbalances and sacroiliac dysfunction can also be the main cause of SIJ pain and low back pain after delivery . Increasing body mass index during pregnancy and after child birth, pre existing back pain before pregnancy and carrying multiple babies are risk factors for SIJ pain during pregnancy and after delivery. There are other factors causing SIJ pain additionally to hypermobility of the joints caused by pregnancy hormones like falling down. The mother might also get this problem, from an activity that gives the area a regular pounding like jogging or if she has one leg longer than the other that could be a cause of SIJ pain. Arthritis can also lead to SIJ pain ( a type that affects the spine called ankylosing spondylitis can damage the SIJ). SIJ pain can also occur when the cartilage over the joint slowly wears away by aging. SIJ pain may occur at any time during pregnancy and becomes more intense as the pregnancy progresses. This pain usually spontaneously resolves within 3 months after delivery. But, in some cases it can become chronic and disabling . SIJ pain could be a dull or sharp. It starts at SIJ but it can move to buttocks, thighs, groin or upper back. Sometimes, standing up trigger the pain and a lot of times the mother feels it only on one side of her lower back. The mother may notice that, it bothers her more in the morning and gets better during the day.There are many choices for treating SIJ pain. The first step is simply to stop any activities that make the mother hurt. The doctor will tell her to lay off any movement or sports that inflame her joints. She may also prescribe some pain drugs. Oral anti-inflammatory medications are often effective in pain relief.

Physiotherapy and exercises that focus on core stability of the trunk and pelvic girdle are considered the main line of treatment for SIJ pain. Sometimes a sacroiliac belt is prescribed to complement the core stability exercises and to give quick pain relief . The core stability exercises are very necessary and will form a large part of the treatment, and in some cases, mobilization (a gentle form of manipulation) of hip, back or pelvis may be used to correct any underlying movement dysfunction Other manual techniques can also be used to treat SIJ pain like muscle energy technique,myofacial release and massage therapy.

ELIGIBILITY:
Inclusion Criteria

1. sacroiliac joint dysfunction
2. severe pain in the sacroiliac joint
3. Age will range from 25 to 35 years old.
4. Body Mass Index: ≤30 kg/m2
5. The type of delivery is a cesarean section.
6. All patients will not receive any medical treatment to relieve pain or decrease inflammation.
7. All patients are not pregnant.

Exclusion Criteria

1. Diabetic mellitus and hypertension
2. Cardiovascular diseases
3. heart diseases
4. Rheumatoid arthritis
5. Cervical spondylosis with radiculopathy or any spinal diseases

(5) leukemia. (6) Deformities in their hands (7) Burns, ulcers, open wounds, or any skin diseases in dominant hands (8) received medications or have been injected with steroids at a tender point.

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — sacroiliac pain in woman postpartum
Enrollment: 40 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale (VAS) | 4 weeks
  This scale will be used by each patient before and after treatment course to estimate the intensity of pain. Visual analogue scale (VAS) is a graphic rating scale with numerical values ranging from 0 to 4, placed equidistantly on a line of 10 cm long drawn horizontally.

CONTACTS AND LOCATIONS:
Locations (1):
- Sadat General Hospital, Cairo, Egypt

REFERENCES:
- [Background] Fiani B, Sekhon M, Doan T, Bowers B, Covarrubias C, Barthelmass M, De Stefano F, Kondilis A. Sacroiliac Joint and Pelvic Dysfunction Due to Symphysiolysis in Postpartum Women. Cureus. 2021 Oct 9;13(10):e18619. doi: 10.7759/cureus.18619. eCollection 2021 Oct. PMID 34786225